CLINICAL TRIAL: NCT06659341
Title: Phase 1 Study of a SOS1 Inhibitor, BAY 3498264, in Combination in Participants With Advanced KRASG12C-mutated Solid Tumors
Brief Title: A Phase I Study of BAY3498264 Given Together With Sotorasib in Participants Who Have Advanced Solid Cancers With Specific Genetic Changes Called KRASG12C Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22676; 2024-513300-34-00 (Registry Identifier: CTIS(EU))
Record Dates: First submitted 2024-10-15; First posted 2024-10-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors Harboring KRAS G12C Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation (Experimental): During dose escalation, at each dose level BAY3498264 monotherapy will be administered for 7 days as a safety run-in, prior to introduction of a combination agent (sotorasib) for 21-day treatment cycles. Intra-participant dose escalation will be implemented: participants will be able to move to a cohort offering a higher dose level of BAY3498264 provided protocol-specified criteria are met.
  Interventions: Drug: BAY3498264
- Backfill cohorts (Experimental): Backfill cohorts may be initiated concurrently with dose escalation cohorts to generate additional safety, PK, and PD data to facilitate the selection of the optimal doses for use in further development.
  Interventions: Drug: BAY3498264
- Exploratory expansion cohorts (Experimental): Exploratory expansion cohorts may be recruited to provide additional safety, PK/PD, and efficacy data.
  Interventions: Drug: BAY3498264

INTERVENTIONS:
Drug: BAY3498264 — Oral

SUMMARY:
Researchers are looking for a better way to treat people who have advanced solid cancers with a KRASG12C mutation.

Sotorasib is a drug that targets cancer cells which contain mutated KRASG12C protein; it can stop the cancer cells from growing and can lead to their death. Sotorasib is already approved to be used by doctors. However, when sotorasib works, it normally only works for a period of time, after which the cancer starts to grow again, and the patient may need a different treatment.

BAY3498264 is a drug that is currently under development. It is expected to prevent the activity of a protein called son of sevenless 1 (SOS1). The SOS1 protein works together with KRAS; by blocking the activity of SOS1 with BAY3498264, it is hoped that the benefit offered by treatment with sotorasib may be increased - for example, resulting in a longer or deeper response.

The main purpose of this first-in-human study is to learn how safe BAY3498264 is when given together with sotorasib and what is the maximum dose of BAY3498264 that can be safely given to participants together with sotorasib.

During the study, participants will receive the following treatments:

* BAY3498264: participants will first receive BAY3498264 alone for seven days and then BAY3498264 in combination with sotorasib. These combination treatments will be given in cycles, each lasting 21 days.
* Sotorasib: participants will receive a standard, approved dose of Sotorasib once every day with BAY3498264.

The treatment will continue for as long as participants benefit from it without any severe medical problems or until they or their doctor decide to stop the treatment, or until their cancer starts to grow again despite the treatment (also called 'progression').

This study has 3 parts, the dose escalation part, the backfill part and the expansion part.

During the study, researchers will collect blood, urine, and take imaging scans like CT, PET, MRI, and X-rays, and examine the participants' heart health using an electrocardiogram (ECG). Participants' health is monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor malignancy with documented KRAS^G12C mutation as assessed by an appropriately accredited laboratory.
* Documented disease progression after treatment with at least 1 prior standard of care (SoC) systemic therapy other than a G12C inhibitor for locally advanced or metastatic disease, and with no further standard treatment options available, or when standard treatment options are not acceptable and this study is a reasonable option.

  * Participants whose access to SoC therapies is limited due to regional access, refusal, intolerance, or eligibility may participate.
  * Prior G12C inhibitor treatment is permitted. Participants receiving prior G12C inhibitor therapy must have documented disease progression after treatment, or have discontinued that treatment due to intolerance.
* Adequate archival formalin-fixed paraffin-embedded tumor tissue available (preferably no older than 6 months, obtained after the last targeted therapy). If archival material is not available, a fresh tumor biopsy should ideally be obtained if safe and feasible.
* Eastern Cooperative Oncology Group (ECOG) of 0 to 2 and life expectancy of at least 12 weeks.

Exclusion Criteria:

- Active central nervous system (CNS) tumors including metastatic brain disease, at the time of screening.

1. 'Active' is defined as untreated brain lesions (new or progressing) or symptomatic brain lesions (as determined by the investigator).
2. Participants who have received treatment (e.g. surgery or radiotherapy) for brain metastases ending at least 4 weeks before the start of study intervention may be eligible if, at the point of study entry:

i. their condition is considered stable by the investigator. ii. they have no residual neurological symptoms (Grade >2). iii. a follow-up Magnetic resonance imaging (MRI) scan during the screening period shows no progression or new lesions.

iv. they do not need systemic corticosteroids to treat symptoms of brain metastasis.

* Any grade active pneumonitis or interstitial lung disease (ILD), or past medical history of:

  1. Grade ≥2 ILD,
  2. Drug-induced ILD,
  3. Radiation pneumonitis that required steroid treatment within the last 12 months.
* Additional malignancy within the past 3 years, except for basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder tumors, localized prostate cancer or other tumors that in the opinion of the investigator, in agreement with the Sponsor, are considered cured or not immediately life-threatening, and will not interfere with the scientific goals of this study.
* Any positive test result for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating the presence of virus.

  * Active HBV (chronic or acute; defined as having a known positive HBsAg test at the time of screening) except for participants on antiviral therapy for HBV with an undetectable or low viral load.
  * Participants with past HBV infection or resolved HBV infection (defined as the presence of HBcAb and absence of HBsAg) are eligible if HBV DNA is negative.
  * Participants positive for HCV antibody unless polymerase chain reaction is negative for HCV RNA. Any prior antiviral therapy must be completed at least 28 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-03-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) categorized by severity. | 30-35 days after the last dose
Maximum tolerated dose (MTD) or Maximum administered dose (MAD) of BAY 3498264 in combination with sotorasib. | Approximate 3 years
Number of participants with Dose-limiting toxicity (DLTs) during the DLT observation period categorized by severity. | DLT evaluation period (Cycle 1) includes 28 days
Maximum observed drug concentration in plasma (Cmax) of the respective dosing interval of BAY3498264 after single dose and multiple dose administrations. | Multiple time points: Cycle 1 28-day cycle followed by 21-day treatment cycles
Area under the concentration vs. time curve (AUC) of the respective dosing interval of BAY3498264 after single dose and multiple dose administrations. | Multiple time points: Cycle 1 28-day cycle followed by 21-day treatment cycles

SECONDARY OUTCOMES:
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) by investigator assessment. | Every 6 weeks (±7 days) for the first 36 weeks and every 9 weeks (± 7 days) thereafter until radiological disease progression (PD) occurs
Recommended dose(s) and schedule(s) of BAY 3498264 to be used in combination with sotorasib for further development stages. | Approximate 3 years

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (3):
  - Border Medical oncology - Albury Wodonga Regional Cancer Centre, Albury, New South Wales
  - Macquarie University Hospital - Oncology Department, Macquarie Park, New South Wales
  - Peninsula and Southeast Oncology, Frankston, Victoria
- Rigshospitalet - Kræftbehandling, Copenhagen OE, Denmark
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Rome, Lazio
  - Gruppo Humanitas - Humanitas Research Hospital - Cancer Center, Rozzano
- Spain (2):
  - Institut Catala D'oncologia | Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall D Hebron | Oncologia, Barcelona
- United Kingdom (2):
  - The Christie NHS Foundation Trust - Christie Hospital, Manchester, Greater Manchester
  - The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital (RMH) - Sutton, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.